CLINICAL TRIAL: NCT02103361
Title: Stelara® and Tremfya® Pregnancy Exposure Registry: OTIS Autoimmune Diseases in Pregnancy Project
Brief Title: Stelara and Tremfya Pregnancy Exposure Registry OTIS Autoimmune Diseases in Pregnancy Project
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: The Organization of Teratology Information Specialists (Other); Janssen Biotech, Inc. (Industry)
Responsible Party: Principal Investigator, Christina Chambers, Professor, Co-Director Center for Promotion of Maternal Health and Infant Development, University of California, San Diego
Other Study IDs: CNTO1275PSO4037
Record Dates: First submitted 2014-02-13; First posted 2014-04-03 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Psoriasis; Pregnancy; Psoriatic Arthritis; Crohn Disease
Keywords: autoimmune disease; pregnancy; psoriasis; Stelara; ustekinumab; birth outcome; malformation; birth defect; psoriatic arthritis; Crohn's Disease; Tremfya; guselkumab
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Crohn Disease; Autoimmune Diseases; Congenital Abnormalities | interventions — Ustekinumab; guselkumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stelara (ustekinumab) exposed: Stelara (ustekinumab)-exposed pregnant women (this group is now closed to recruitment)
  Interventions: Drug: Ustekinumab
- Tremfya (guselkumab) exposed: Tremfya (guselkumab-exposed pregnant women
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Ustekinumab
  Other Names: Stelara
  Groups: Stelara (ustekinumab) exposed
Drug: Guselkumab
  Other Names: Tremfya
  Groups: Tremfya (guselkumab) exposed

SUMMARY:
The purpose of the OTIS Autoimmune Diseases in Pregnancy Study is to monitor planned and unplanned pregnancies exposed to certain medications, to evaluate the possible teratogenic effect of these medications and to follow live born infants for one year after birth. With respect to fetal outcome, it is important to evaluate the spectrum of outcomes that may be relevant to a medication exposure during pregnancy, and these include both easily recognizable defects which are visible at birth, as well as more subtle or delayed defects that may not be readily identifiable without special expertise and observation beyond the newborn period.

DETAILED DESCRIPTION:
The purpose of the Stelara and Tremfya Pregnancy Exposure Registry OTIS Autoimmune Diseases in Pregnancy Project is to follow pregnant women or women who have delivered a baby, who have been treated with Stelara or Tremfya within 3 months of their last menstrual period (LMP) or during pregnancy to evaluate the possible effect of this medication on the pregnancy outcome including child development and growth up to one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of an exposure to Stelara (ustekinumab) or Tremfya (guselkumab) during pregnancy or within 3 months prior to the first day of the last menstrual period (LMP) for any number of days, at any time, at any dose, and at any time until completion of pregnancy.
* Documentation of gestational timing of the exposure to Stelara (ustekinumab) or Tremfya (guselkumab)

Exclusion Criteria:

* Women who have not have an exposure to Stelara (ustekinumab) or Tremfya (guselkumab) during pregnancy or within 3 months of the first day of the last menstrual period.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women who have had exposure to Stelara (ustekinumab) or Tremfya (guselkumab) within 3 months of the last menstrual period, or anytime during pregnancy, and who reside in the U.S. or Canada.
  The Stelara (ustekinumab) exposed group completed enrollment as of September 2019. The Tremfya (guselkumab) remains open to recruitment.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Major structural malformations | From 3 months prior to the first day of the last menstrual period and up to one year of age
  The primary objective of the study is to evaluate the effect of certain medications when used in the first trimester of pregnancy with respect to major structural birth defects.

SECONDARY OUTCOMES:
Minor Congenital Structural Malformations | At dysmorphological exam which will occur at one time point between birth and one year of age
  One secondary objective of the study is to evaluate the effects of certain medications when used in the first trimester of pregnancy with respect to potential minor malformations.

OTHER OUTCOMES:
Spontaneous abortions | From 3 months prior to the first day of the last menstrual period until the day of delivery
  Rate of spontaneous abortions
Infant follow-up, growth | Birth to one year of age
  Pre- and post-natal fetal and infant growth, small for gestational age, and preterm delivery
Stillbirths | From 3 months prior to the first day of the last menstrual period until the day of delivery
  Rate of stillbirth
Infant follow-up, Immune system development | Birth to 1 year of age
  Health and development including effects to the immune system development.
Preterm delivery | Birth
  Rate of preterm delivery

CONTACTS AND LOCATIONS:
Overall Officials: Christina Chambers, PhD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- See also: Official research website of the Organization of Teratology Information Specialists, Studies coordinated at the University of California, San Diego — https://mothertobaby.org/pregnancy-studies/